CLINICAL TRIAL: NCT02190058
Title: A PHASE I, DOUBLE-BLIND, RANDOMISED, PLACEBO-CONTROLLED, MULTIPLE-DOSE STUDY TO ASSESS SAFETY, TOLERABILITY AND PHARMACOKINETICS OF DS-1971A IN HEALTHY MALE SUBJECTS
Brief Title: Multiple Dose Study of DS-1971a
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DS1971-A-E102
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2015-01

CONDITIONS: Healthy
Keywords: safety; pharmacokinetics; DS-1971a
MeSH Terms: interventions — DS-1971a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DS-1971a (Experimental): DS-1971a suspension, up to 4650mg/day
  Interventions: Drug: DS-1971a
- placebo (Placebo Comparator): matching DS-1971a suspension
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: DS-1971a — suspension
  Arms: DS-1971a
Drug: placebo — placebo matching DS-1971a
  Arms: placebo

SUMMARY:
This is a randomised, double-blind, placebo-controlled multiple dose study designed to explore the safety, tolerability and PK of DS-1971a following oral administration over 14 days to healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 18-55 years.
* A body mass index (BMI) in the range 18-30 kg/m2, inclusive, and weighing between 50 and 100 kg at screening.
* Willing to comply with all study restrictions, including the use of contraception, concomitant medication, and dietary and lifestyle restrictions.
* Sufficient intelligence to understand the nature of the study and any hazards of participating in it. Ability to communicate satisfactorily with the Investigator and to participate in, and comply with requirements of, the entire study.
* Have given written consent to participate in the study after reading the ICF, and after having the opportunity to discuss the study with the Investigator or his delegate.
* Have given written consent to have his data entered into The Over-volunteering Prevention System.

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, ECG findings, or laboratory values that could interfere with the objectives of the study or compromise the safety of the subject.
* Presence or history of acute or chronic illness, including (but not limited to) liver or kidney disease, hypertension, seizures, or any known impairment of endocrine, or other specific body-organ dysfunction.
* History of serious reaction to any medicine.
* Presence or history of malignant disease.
* Acute or chronic infectious disease, including human immunodeficiency virus (HIV), hepatitis B virus (HBV) or C virus (HCV) infection.
* Surgery (eg stomach bypass) or medical condition that might affect how the body handles or absorbs medicines.
* Significant illness within 4 weeks before the first dose of study medication.
* Participation in another clinical study of a new chemical entity or a prescription medicine within the previous 3 months, or unwilling to abstain from participating in other clinical trials during the study and for 3 months after receipt of study medication.
* Participation in another clinical study with DS 1971a.
* Abnormal ECG waveform morphology at screening that would preclude accurate measurement of the QT interval duration.
* Corrected QT interval (Fridericia's formula) (QTcF) interval duration > 430 msec, obtained as an average from the measurements on duplicate screening ECGs.
* Estimated glomerular filtration rate (eGFR) < 80 mL/min/1.73m2 (based on Modification of Diet in Renal Disease [MDRD] equation) or an absolute creatinine value outside the normal range.
* Use of any prescription or over the counter (OTC) medications, or herbal remedies (such as St John's wort), known to be strong inhibitors or strong inducers of cytochrome (CYP) enzymes (also known as CYP P450 enzymes) during the 30 days before the first dose of study medication; use of any other prescription or OTC medicine (with the exception of acetaminophen (paracetamol)), including dietary supplements or herbal remedies, during the 7 days before the dose of study medication.
* Consumption of certain foods or beverages before the first dose and throughout the study period.
* Loss of more than 400 mL blood or donation of blood, plasma, platelets, or any other blood components during the 3 months before the first dose of study medication, or unwilling to abstain from doing so during the study and for 3 months after receipt of study medication.
* Abuse of drugs or alcohol during the 2 years before the first dose of study medication, or intake of more than 21 units of alcohol weekly.
* Use of tobacco products or nicotine-containing products during the 3 months before the first dose of study medication and during the study.
* Evidence of drug or alcohol abuse at screening or admission.
* Likely possibility that the volunteer will not cooperate with the requirements of the protocol.
* Objection by GP to the volunteer entering the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
adverse events | up to 2 months
  To assess the safety and tolerability of repeated oral doses of DS-1971a in healthy male subjects the number, severity, and frequency of adverse events will be recorded from enrollment through discharge from study, up to 2 months.

SECONDARY OUTCOMES:
characterise the plasma pharmacokinetics AUC (area under curve) | Day 1 through Day 17
  To characterise the plasma pharmacokinetics (PK) of DS-1971a in healthy male subjects receiving repeated oral doses.
  plasma concentrations of DS 1971a, and derived PK parameters: AUC (area under curve); Cmax (maximum concentration); Tmax (time of maximum concentration), T½ (terminal half-life), CL/F; Vss/F
characterise the plasma pharmacokinetics Cmax (maximum concentration) | Day 1 through Day 17
  To characterise the plasma pharmacokinetics (PK) of DS-1971a in healthy male subjects receiving repeated oral doses.
  plasma concentrations of DS 1971a, and derived PK parameters: AUC (area under curve); Cmax (maximum concentration); Tmax (time of maximum concentration), T½ (terminal half-life), CL/F; Vss/F
characterise the plasma pharmacokinetics Tmax (time of maximum concentration) | Day 1 through Day 17
  To characterise the plasma pharmacokinetics (PK) of DS-1971a in healthy male subjects receiving repeated oral doses.
  plasma concentrations of DS 1971a, and derived PK parameters: AUC (area under curve); Cmax (maximum concentration); Tmax (time of maximum concentration), T½ (terminal half-life), CL/F; Vss/F
characterise the plasma pharmacokinetics T½ (terminal half-life) | Day 1 through Day 17
  To characterise the plasma pharmacokinetics (PK) of DS-1971a in healthy male subjects receiving repeated oral doses.
  plasma concentrations of DS 1971a, and derived PK parameters: AUC (area under curve); Cmax (maximum concentration); Tmax (time of maximum concentration), T½ (terminal half-life), CL/F; Vss/F
characterise the plasma pharmacokinetics CL/F (apparent oral clearance) | Day 1 through Day 17
  To characterise the plasma pharmacokinetics (PK) of DS-1971a in healthy male subjects receiving repeated oral doses.
  plasma concentrations of DS 1971a, and derived PK parameters: AUC (area under curve); Cmax (maximum concentration); Tmax (time of maximum concentration), T½ (terminal half-life), CL/F (apparent oral clearance); Vss/F
characterise the plasma pharmacokinetics Vss/F (apparent volume of distribution) | Day 1 through Day 17
  To characterise the plasma pharmacokinetics (PK) of DS-1971a in healthy male subjects receiving repeated oral doses.
  plasma concentrations of DS 1971a, and derived PK parameters: AUC (area under curve); Cmax (maximum concentration); Tmax (time of maximum concentration), T½ (terminal half-life), CL/F (apparent oral clearance); Vss/F (apparent volume of distribution).

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research Ltd., London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/